CLINICAL TRIAL: NCT02641691
Title: Non-Operative Radiation Management of Adenocarcinoma of the Lower Rectum (NORMAL-R)
Brief Title: Non-Operative Radiation Management of Adenocarcinoma of the Lower Rectum
Acronym: NORMAL-R
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201512140
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cancer of Rectum; Cancer of the Rectum; Neoplasm, Rectum; Rectal Cancer; Rectum Cancer; Rectum Neoplasms; Adenocarcinoma of the Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU (Experimental): * Radiotherapy will consist of five fractions, delivered once daily, to a total dose of 25Gy at 5 Gy per fraction.
  * An optional concomitant boost may be delivered to the primary tumor of 1-2 Gy per day (30-35 Gy to tumor total). If a boost is given then the maximum allowed dose to small bowel is 25 Gy.
  * Chemotherapy should begin two weeks (9-12 working days) after completion of radiotherapy.
  * Oxaliplatin will be given intravenous (IV) over 2 hours on Day 1 every 14 days for a maximum of 8 cycles.
  * Leucovorin will be given IV over 2 hours on Day 1 every 14 days for a maximum of 8 cycles.
  * 5-FU bolus will given IV push on Day 1 every 14 days for a maximum of 8 cycles.
  * 5-FU infusion will be given continuous IV on Day 1 over 46 hours every 14 days for a maximum of 8 cycles
  * Alternatively, capecitabine/oxaliplatin (CAPE PO 1000 mg/m2 BID days 1-14 Q21 days, oxaliplatin IV 130 mg/m2 IV Q21 days on day 1) x 5 cycles over 15 weeks may be administered instead of FOLFOX
  Interventions: Radiation: Radiation; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Radiation: Radiation
Drug: Oxaliplatin
  Other Names: Eloxatin®
Drug: Leucovorin
  Other Names: Wellcovorin; citrovorum factor; folinic acid; 5-formyl tetrahydrofolate
Drug: Fluorouracil
  Other Names: 5-Fluorouracil; 5-FU

SUMMARY:
The purpose of this research study is to look at how tumors responds to a short course of radiation (5 days) followed by 8 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of biopsy proven stage I-IIIB (cT1-3, N0-1, M0) adenocarcinoma of the rectum; staging must also be based on multidisciplinary evaluation including MRI and/or endorectal ultrasound
* Tumor ≤ 12 cm from anal verge as determined by MRI or endoscopy a
* ECOG performance status 0-2
* At least 18 years of age
* Adequate bone marrow function defined as:

  * ANC > 1,500 cells/mm3
  * Hgb > 8 g/dl
  * platelets >100,000 cells/mm3
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* No clinically detectable (MR, endoscopy or DRE) tumor present
* Prior radiation therapy, chemotherapy or extirpative surgery for rectal cancer.
* Any evidence of disease from another malignancy or history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix). Patients with history of prostate cancer treated without radiotherapy and no evidence of disease are eligible.
* Currently receiving any investigational agents.
* A history of allergic reaction attributed to compounds of similar chemical or biologic composition to 5FU, oxaliplatin, or leucovorin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study entry.
* Known HIV-positivity and on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with the study drugs. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Pedersen K, Olsen JR, Mutch MG, Chin RI, Glasgow SC, Wise PE, Silviera ML, Tan BR, Wang-Gillam A, Lim KH, Suresh R, Amin M, Huang Y, Henke LE, Park H, Ciorba MA, Badiyan S, Parikh PJ, Roach MC, Hunt SR. Nonoperative Rectal Cancer Management With Short-Course Radiation Followed by Chemotherapy: A Nonrandomized Control Trial. Clin Colorectal Cancer. 2021 Sep;20(3):e185-e193. doi: 10.1016/j.clcc.2021.03.003. Epub 2021 Apr 7. PMID 34001462
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 56.5 [38 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: * Criteria for complete clinical response:
    * No residual gross tumor at procto/sigmoidoscopy, or only erythematous scar or ulcer
    * No radiographic evidence of tumor on DRE
    * Substantial downsizing on MRI
    * No suspicious mesorectal lymph nodes on MRI
    * Negative biopsy from scar, ulcer, or former tumor site (if necessary according to surgeon's judgment)
  * Criteria for no significant clinical response:
    * Residual disease by DRE, endoscopy or MR.
    * Increase in primary tumor size upon clinical exam or imaging
    * Any new lesions
Time Frame: 1 year
Population: 1 participant was not evaluable for this outcome measure as they were removed for an adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 19
Participants | 12

2. Secondary Outcome: Prospective Patient Reported Outcomes as Measured by FACT-C Questionnaire
Description: -The FACT-C questionnaire is broken down into physical well-being, social/family well-being, emotional well-being, and functional well-being. The answers range from 0 (not at all) to 4 (very much).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- 0=Not at All; 1=A Little Bit; 2=Somewhat; 3=Quite a Bit; 4=Very Much: -Participant is asked about specific well-being in the past 7 days
- Prefer Not to Answer/No Answer/No: -Participant did not answer question about well-being
Arm/Group | 0=Not at All | 1=A Little Bit | 2=Somewhat | 3=Quite a Bit | 4=Very Much | Prefer Not to Answer/No Answer/No
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
Participants
  I have a lack of energy | 9 | 3 | 6 | 2 | 0 | 0
  I have nausea | 19 | 0 | 1 | 0 | 0 | 0
  Because of my physical condition, I have trouble meeting the needs of my family | 17 | 2 | 1 | 0 | 0 | 0
  I have pain | 11 | 6 | 2 | 1 | 0 | 0
  I am bothered by side effects of treatment | 19 | 0 | 0 | 0 | 0 | 1
  I feel ill | 19 | 0 | 1 | 0 | 0 | 0
  I am forced to spend time in bed | 17 | 1 | 1 | 0 | 0 | 1
  I feel close to my friends | 0 | 0 | 1 | 1 | 18 | 0
  I get emotional support from my family | 0 | 0 | 0 | 0 | 20 | 0
  I get support from my friends | 0 | 0 | 0 | 1 | 19 | 0
  My family has accepted my illness | 0 | 0 | 0 | 2 | 18 | 0
  I am satisfied with family communication about my illness | 0 | 0 | 0 | 1 | 19 | 0
  I feel close to my partner (or the person who is my main support) | 0 | 0 | 1 | 0 | 19 | 0
  I am satisfied with my sex life | 0 | 1 | 6 | 1 | 8 | 4
  I feel sad | 8 | 8 | 4 | 0 | 0 | 0
  I am satisfied with how I am coping with my illness | 2 | 2 | 4 | 5 | 7 | 0
  I am losing hope in the fight against my illness | 19 | 1 | 0 | 0 | 0 | 0
  I feel nervous | 6 | 4 | 4 | 4 | 2 | 0
  I worry about dying | 12 | 4 | 2 | 2 | 0 | 0
  I worry that my condition will get worse | 2 | 9 | 5 | 4 | 0 | 0
  I am able to work (include work at home) | 0 | 1 | 3 | 4 | 12 | 0
  My work (include work at home) is fulfilling | 0 | 0 | 5 | 3 | 11 | 1
  I am able to enjoy life | 0 | 0 | 2 | 3 | 15 | 0
  I have accepted my illness | 0 | 0 | 2 | 6 | 12 | 0
  I am sleeping well | 2 | 0 | 6 | 6 | 6 | 0
  I am enjoying the things I usually do for fun | 0 | 0 | 4 | 7 | 9 | 0
  I am content with the quality of my life right now | 0 | 1 | 6 | 6 | 7 | 0
  I have swelling or cramps in my stomach area | 14 | 5 | 0 | 0 | 1 | 0
  I am losing weight | 10 | 5 | 2 | 3 | 0 | 0
  I have control of my bowels | 1 | 0 | 5 | 3 | 11 | 0
  I can digest my food well | 0 | 0 | 2 | 4 | 13 | 1
  I have diarrhea (diarrhoea) | 9 | 5 | 4 | 0 | 2 | 0
  I have a good appetite | 1 | 0 | 0 | 6 | 13 | 0
  I like the appearance of my body | 0 | 2 | 4 | 8 | 6 | 0
  I am embarrassed by my ostomy appliance | 0 | 0 | 0 | 0 | 0 | 20
  Caring for my ostomy appliance is difficult | 0 | 0 | 0 | 0 | 0 | 20

3. Secondary Outcome: Prospective Patient Reported Outcomes as Measured by FACT-C Questionnaire
Description: as for outcome 2
Time Frame: Completion of chemoradiation (approximately 112 days)
Population: One participant was not evaluable for this outcome measure because they did not complete chemoradiation.
Measure: Count of Participants; unit: Participants
Arm/Group | 0=Not at All | 1=A Little Bit | 2=Somewhat | 3=Quite a Bit | 4=Very Much | Prefer Not to Answer/No Answer/No
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19
Participants
  I have a lack of energy | 3 | 3 | 11 | 2 | 0 | 0
  I have nausea | 16 | 3 | 0 | 0 | 0 | 0
  Because of my physical condition, I have trouble meeting the needs of my family | 8 | 8 | 2 | 0 | 1 | 0
  I have pain | 11 | 3 | 4 | 0 | 0 | 1
  I am bothered by side effects of treatment | 6 | 7 | 3 | 2 | 1 | 0
  I feel ill | 16 | 2 | 0 | 0 | 0 | 1
  I am forced to spend time in bed | 13 | 6 | 0 | 0 | 0 | 0
  I feel close to my friends | 0 | 1 | 1 | 3 | 14 | 0
  I get emotional support from my family | 0 | 1 | 1 | 2 | 15 | 0
  I get support from my friends | 1 | 0 | 1 | 1 | 16 | 0
  My family has accepted my illness | 1 | 0 | 1 | 3 | 14 | 0
  I am satisfied with family communication about my illness | 1 | 0 | 2 | 2 | 14 | 0
  I feel close to my partner (or the person who is my main support) | 0 | 0 | 2 | 0 | 17 | 0
  I am satisfied with my sex life | 1 | 1 | 8 | 1 | 5 | 3
  I feel sad | 10 | 5 | 3 | 1 | 0 | 0
  I am satisfied with how I am coping with my illness | 3 | 0 | 4 | 8 | 4 | 0
  I am losing hope in the fight against my illness | 16 | 1 | 2 | 0 | 0 | 0
  I feel nervous | 5 | 11 | 3 | 0 | 0 | 0
  I worry about dying | 12 | 6 | 0 | 1 | 0 | 0
  I worry that my condition will get worse | 4 | 11 | 3 | 1 | 0 | 0
  I am able to work (include work at home) | 1 | 4 | 3 | 3 | 8 | 0
  My work (include work at home) is fulfilling | 0 | 4 | 5 | 2 | 8 | 0
  I am able to enjoy life | 0 | 2 | 3 | 7 | 7 | 0
  I have accepted my illness | 1 | 2 | 1 | 6 | 9 | 0
  I am sleeping well | 0 | 2 | 3 | 6 | 7 | 1
  I am enjoying the things I usually do for fun | 0 | 3 | 4 | 6 | 6 | 0
  I am content with the quality of my life right now | 0 | 2 | 6 | 5 | 6 | 0
  I have swelling or cramps in my stomach area | 13 | 4 | 1 | 1 | 0 | 0
  I am losing weight | 11 | 6 | 1 | 0 | 0 | 1
  I have control of my bowels | 1 | 4 | 6 | 4 | 4 | 0
  I can digest my food well | 0 | 2 | 3 | 3 | 10 | 1
  I have diarrhea (diarrhoea) | 4 | 10 | 2 | 2 | 1 | 0
  I have a good appetite | 1 | 1 | 5 | 7 | 4 | 1
  I like the appearance of my body | 2 | 3 | 8 | 3 | 3 | 0
  I am embarrassed by my ostomy appliance | 1 | 0 | 0 | 0 | 0 | 18
  Caring for my ostomy appliance is difficult | 1 | 0 | 0 | 0 | 0 | 18

4. Secondary Outcome: Prospective Patient Reported Outcomes as Measured by FACT-C Questionnaire
Description: as for outcome 2
Time Frame: 10-14 months after chemoradiation (approximately 16-20 months)
Population: One participant was not evaluable for this outcome measure because they did not complete chemoradiation. One participant was not evaluable for this outcome measure because they expired prior to this timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | 0=Not at All | 1=A Little Bit | 2=Somewhat | 3=Quite a Bit | 4=Very Much | Prefer Not to Answer/No Answer/No
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18
Participants
  I have a lack of energy | 4 | 5 | 5 | 4 | 0 | 0
  I have nausea | 17 | 0 | 1 | 0 | 0 | 0
  Because of my physical condition, I have trouble meeting the needs of my family | 10 | 4 | 4 | 0 | 0 | 0
  I have pain | 9 | 5 | 3 | 0 | 1 | 0
  I am bothered by side effects of treatment | 5 | 2 | 6 | 3 | 2 | 0
  I feel ill | 15 | 2 | 1 | 0 | 0 | 0
  I am forced to spend time in bed | 14 | 2 | 1 | 1 | 0 | 0
  I feel close to my friends | 0 | 0 | 2 | 4 | 12 | 0
  I get emotional support from my family | 0 | 0 | 1 | 2 | 15 | 0
  I get support from my friends | 0 | 0 | 2 | 2 | 13 | 1
  My family has accepted my illness | 0 | 0 | 2 | 2 | 14 | 0
  I am satisfied with family communication about my illness | 0 | 0 | 1 | 1 | 15 | 1
  I feel close to my partner (or the person who is my main support) | 0 | 0 | 2 | 1 | 15 | 0
  I am satisfied with my sex life | 5 | 0 | 2 | 2 | 4 | 5
  I feel sad | 9 | 6 | 3 | 0 | 0 | 0
  I am satisfied with how I am coping with my illness | 3 | 0 | 4 | 4 | 7 | 0
  I am losing hope in the fight against my illness | 15 | 1 | 1 | 0 | 1 | 0
  I feel nervous | 6 | 6 | 4 | 1 | 1 | 0
  I worry about dying | 10 | 5 | 2 | 1 | 0 | 0
  I worry that my condition will get worse | 5 | 7 | 5 | 1 | 0 | 0
  I am able to work (include work at home) | 1 | 2 | 3 | 3 | 9 | 0
  My work (include work at home) is fulfilling | 1 | 0 | 6 | 2 | 9 | 0
  I am able to enjoy life | 0 | 1 | 5 | 5 | 7 | 0
  I have accepted my illness | 0 | 0 | 5 | 5 | 7 | 1
  I am sleeping well | 1 | 1 | 4 | 5 | 6 | 1
  I am enjoying the things I usually do for fun | 0 | 4 | 4 | 6 | 3 | 1
  I am content with the quality of my life right now | 0 | 5 | 5 | 3 | 4 | 1
  I have swelling or cramps in my stomach area | 12 | 1 | 2 | 2 | 1 | 0
  I am losing weight | 15 | 2 | 0 | 0 | 1 | 0
  I have control of my bowels | 2 | 2 | 7 | 5 | 2 | 0
  I can digest my food well | 0 | 1 | 5 | 2 | 10 | 0
  I have diarrhea (diarrhoea) | 6 | 6 | 2 | 2 | 2 | 0
  I have a good appetite | 1 | 0 | 3 | 4 | 10 | 0
  I like the appearance of my body | 3 | 2 | 8 | 2 | 3 | 0
  I am embarrassed by my ostomy appliance | 1 | 0 | 1 | 0 | 1 | 15
  Caring for my ostomy appliance is difficult | 1 | 2 | 0 | 0 | 0 | 15

5. Secondary Outcome: Number of Any Grade 3 or Higher Toxicities
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: From start of radiation treatment through 30 days after completion of treatment (approximately 18 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 20
Participants
  Anemia | 2
  Febrile neutropenia | 2
  Cardiac arrest | 1
  Myocardial infarction | 1
  Ventricular fibrillation | 1
  Abdominal pain | 1
  Diarrhea | 3
  Pancreatitis | 1
  Fever | 1
  Cholectystitis | 1
  Lung infection | 1
  Fall | 1
  Activated partial thromboplastin time prolonged | 1
  Aspartate aminotransferase increased | 1
  Cardiac troponin I increased | 1
  Cardiac troponin T increased | 1
  Lymphocyte count decreased | 3
  Neutrophil count decreased | 5
  White blood cell decreased | 2
  Dehydration | 2
  Hyperglycemia | 1
  Hypokalemia | 2
  Hyponatremia | 2
  Generalized muscle weakness | 1
  Peripheral sensory neuropathy | 2
  Syncope | 1
  Respiratory failure | 1
  Aspiration | 1
  Dyspnea | 2
  Hypoxia | 1
  Palmar-plantar erythrodysesthesia syndrome | 1
  Cellulitis | 1
  Hypertension | 1
  Hypotension | 2
  Thromboembolic event | 1

6. Secondary Outcome: Number of Post Chemotherapy Grade 3 or Higher Toxicities
Description: as for outcome 5
Time Frame: Post-chemotherapy through 1 year follow-up (approximately 1 year and 4 months)
Population: One participant was not evaluable for this outcome measure because they did not complete chemoradiation.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 19
Participants
  Anemia | 2
  Febrile neutropenia | 2
  Cardiac arrest | 1
  Myocardial infarction | 1
  Ventricular fibrillation | 1
  Abdominal pain | 1
  Diarrhea | 3
  Fever | 2
  Cholecystitis | 1
  Lung infection | 1
  Activated partial thromboplastin time prolonged | 1
  Aspartate aminotransferase increased | 1
  Cardiac troponin I increased | 1
  Cardiac troponin T increased | 1
  Lymphocyte count decreased | 3
  Neutrophil count decreased | 5
  White blood cell count decreased | 2
  Dehydration | 1
  Hyperglycemia | 1
  Hypokalemia | 2
  Hyponatremia | 2
  Generalized muscle weakness | 1
  Peripheral sensory neuropathy | 2
  Syncope | 1
  Respiratory failure | 1
  Aspiration | 1
  Dyspnea | 1
  Hypoxia | 1
  Cellulitis | 1
  Hypotension | 1
  Thromboembolic event | 1

7. Secondary Outcome: Quality of Anorectal Function as Measured by the FACT-C Questionnaire
Description: -The FACT-C questionnaire has 2 statements about anorectal function and the participant answers 0 (not at all) to 4 (very much)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 0=Not at All | 1=A Little Bit | 2=Somewhat | 3=Quite a Bit | 4=Very Much
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
Participants
  I have control of my bowels | 1 | 0 | 5 | 3 | 11
  I have diarrhea (diarrhoea) | 9 | 5 | 4 | 0 | 2

8. Secondary Outcome: Quality of Anorectal Function as Measured by the FACT-C Questionnaire
Description: as for outcome 7
Time Frame: Completion of chemoradiation (approximately 112 days)
Population: One participant was not evaluable for this outcome measure because they did not complete chemoradiation.
Measure: Count of Participants; unit: Participants
Arm/Group | 0=Not at All | 1=A Little Bit | 2=Somewhat | 3=Quite a Bit | 4=Very Much
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19
Participants
  I have control of my bowels | 1 | 4 | 6 | 4 | 4
  I have diarrhea (diarrhoea) | 4 | 10 | 2 | 2 | 1

9. Secondary Outcome: Quality of Anorectal Function as Measured by the FACT-C Questionnaire
Description: as for outcome 7
Time Frame: 10-14 months after chemoradiation (approximately 16-20 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | 0=Not at All | 1=A Little Bit | 2=Somewhat | 3=Quite a Bit | 4=Very Much
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
Participants
  I have control of my bowels | 2 | 2 | 7 | 5 | 2
  I have diarrhea (diarrhoea) | 6 | 6 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment until 1 year post start of radiation therapy (approximately 1 year and 4 months).
Arm/Group | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU (N=20)
Dehydration (Metabolism and nutrition disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Syncope (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 1
Hypotension (Vascular disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Radiation/Oxaliplatin/Leucovorin/5-FU (N=20)
Anemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Aspartate aminotransferase (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
Cardiac troponin T increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Leg pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (General disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 — Tingling in fingers
Cold sensitivity (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Bottom of feet felt sun burnt (Skin and subcutaneous tissue disorders) | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02641691/Prot_SAP_000.pdf